CLINICAL TRIAL: NCT05322707
Title: Multicenter Randomized Parallel-Group 6-Week Treatment Clinical Study to Assess BE of Budesonide 80 μg and Formoterol Fumarate Dihydrate 4.5 μg Inhalation Product in Comparison With Reference Product, Symbicort® in Adult Asthma Patients
Brief Title: BE Study Budesonide 80 μg and Formoterol Fumarate Dihydrate 4.5 μg Inhalation Product in Asthma Patient
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cipla Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRD/20
Record Dates: First submitted 2022-03-31; First posted 2022-04-12 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Budesonide 80 μg and Formoterol Fumarate Dihydrate 4.5 μg (Experimental): Inhalation Aerosol, 2 actuations orally inhaled twice daily
  Interventions: Drug: Budesonide 80 μg and Formoterol Fumarate Dihydrate 4.5 μg
- Symbicort® (Active Comparator): Inhalation Aerosol, 2 actuations orally inhaled twice daily
  Interventions: Drug: Symbicort, 80 Mcg-4.5 Mcg/Inh Inhalation Aerosol
- Placebo for Budesonide 80 μg and Formoterol Fumarate Dihydrate 4.5 μg (Placebo Comparator): Inhalation Aerosol, 2 actuations orally inhaled twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide 80 μg and Formoterol Fumarate Dihydrate 4.5 μg — Inhalation aerosol, 2 actuations orally inhaled twice daily
  Other Names: Test product
  Arms: Budesonide 80 μg and Formoterol Fumarate Dihydrate 4.5 μg
Drug: Symbicort, 80 Mcg-4.5 Mcg/Inh Inhalation Aerosol — Inhalation aerosol, 2 actuations orally inhaled twice daily
  Other Names: RLD
  Arms: Symbicort®
Drug: Placebo — Inhalation aerosol, 2 actuations orally inhaled twice daily
  Other Names: Placebo for Budesonide 80 μg and Formoterol Fumarate Dihydrate 4.5 μg
  Arms: Placebo for Budesonide 80 μg and Formoterol Fumarate Dihydrate 4.5 μg

SUMMARY:
The purpose of the study is to demonstrate the Pharmacodynamic bioequivalence of the test product to the reference product in adult patient with Asthma

DETAILED DESCRIPTION:
This study is to demonstrate the Pharmacodynamic bioequivalence of the test product to the reference product in terms of FEV1 measures at different timepoints in adult patient with Asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who are 18-70 years of age
* Has moderate-to-severe asthma with a pre-bronchodilator FEV1 of ≥45% and <80% of the predicted normal value for the patient after withholding bronchodilators
* Has ≥15% and ≥0.20 L reversibility of FEV1 within 30 minutes following administration of 360 μg of albuterol (pMDI)
* Is stable on current chronic asthma treatment (documented asthma diagnosis and/or prescription for asthma medications) for at least 4 weeks prior to screening visit (Visit 1).
* Has been diagnosed with asthma as defined by the National Asthma Education and Prevention Program (NAEPP 2007) at least 6 months prior to screening
* Adult male or female patients of non-childbearing or of childbearing potential committed to consistent and correct use of an acceptable method of birth control

Exclusion Criteria:

* Has history of life-threatening asthma defined as an asthma episode(s) that required intubation and/or was associated with hypercapnia, respiratory arrest, or hypoxic seizures, asthma related syncopal episode(s), within past 1 year or during run-in period
* Has history of any asthma-related hospitalizations within the past one year prior to screening visit (Visit 1) or during the run-in period
* Has history of any pulmonary disorder other than asthma, including but not limited to: diagnosis of chronic obstructive pulmonary disease (COPD), interstitial lung disease, cystic fibrosis, bronchiectasis, chronic bronchitis, pulmonary hypertension, active pulmonary tuberculosis, or pulmonary carcinoma.
* Has current evidence of bronchopulmonary dysplasia or pulmonary fibrosis
* Has recent respiratory tract infection that is not resolved within 4 weeks of screening and is considered significant in the opinion of the investigator
* Patients who, in the opinion of the investigator, significantly abuse alcohol or drugs, will be excluded.
* Is taking any immunosuppressive medications within 4 weeks prior to the screening and during the study
* Use of systemic or oral corticosteroids within 2 months or intramuscular depot corticosteroid treatment 90 days prior to the screening or during the run-in period for any reason other than asthma.
* Women of childbearing potential who are lactating or pregnant at screening visit, as documented by a positive screening pregnancy test.
* Has previously been randomized in this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1485 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Area under the serial Force Expiration volume1 | From time 0 to 12 hours
  Area under the serial Force Expiration volume1 from time 0 to 12 hours (AUC0-12 hours) on the first day of the treatment
Change in FEV1 from baseline | 6 weeks treatment
  FEV1 measured in the morning prior to the dosing of inhaled medication on the last day of the 6 weeks treatment

SECONDARY OUTCOMES:
Number and Severity of Adverse Events and Serious Adverse Events | 6 weeks treatment
  Assessment of No. of AEs, its severity, and relatedness and SAE.,
Assessment of vital signs: Pulse rate | 6 weeks treatment
  Assessment of vital signs
Number of participants with suspected oral infection performed with an oropharyngeal examination | 6 weeks treatment
  Assessment of physical examination including oropharyngeal examination
Assessment of vital signs: Systolic and diastolic Blood Pressures | 6 weeks treatment
  Assessment of vital signs: Systolic and diastolic Blood Pressures

CONTACTS AND LOCATIONS:
Overall Officials: Orlando Rivero, MD, Principal Investigator — Global Research Solution
Locations (1):
- Velocity Clinical Research, Medford, Oregon, United States

IPD SHARING:
Plan to Share IPD: No